CLINICAL TRIAL: NCT04418700
Title: Effects of the Breath Stacking Technique After Upper Abdominal Surgery: Randomized Controlled Trial
Brief Title: Effects of the Breath Stacking Technique After Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Prof. Dr. Antônio Marcos Vargas da Silva, Principal Investigator, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11041019.0.0000.5346
Record Dates: First submitted 2020-05-21; First posted 2020-06-05 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Abdominal Surgery
Keywords: surgery; abdomen; pulmonary ventilation; physical therapy techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breath Stacking technique (Experimental): The intervention group will receive routine physical therapy associated with the Breath Stacking technique in 2 daily sessions of up to 20 minutes.
  The technique consists of an Instrument composed of a one-way valve coupled to a face mask to promote the accumulation of successive inspiratory volumes.
  Interventions: Device: Breath Stacking
- Routine physical therapy (No Intervention): The control group will receive only routine physical therapy. Routine physiotherapy consists of breathing exercises, using techniques bronchial hygiene and pulmonary reexpansion, and motor physiotherapy through exercise passive, active-assisted or active mobilization, stretching, training activities of daily living, positioning and removal of the bed and guidelines for post-discharge.

INTERVENTIONS:
Device: Breath Stacking — The patients will perform the maneuver through successive inspiratory efforts for 20 s. Subsequently, the expiratory branch will be unobstructed to allow expiration. This maneuver will be repeated 5 times in each series, with intervals of 30 seconds between them. The technique will be performed with the trunk inclined 30º in relation to the horizontal plane, in 3 series, with interval of 2 min completing 15 min of therapy.
  Arms: Breath Stacking technique

SUMMARY:
This study evaluates the effects of the breath stacking technique in patients after upper abdominal surgery. Half of the patients receive routine physical therapy associated with the Breath Stacking technique, while the other half will receive only routine physical therapy.

DETAILED DESCRIPTION:
This randomized controlled study aims to evaluate the effects of the Breath Stacking technique in patients undergoing upper abdominal surgery on clinical, physiological and cardiopulmonary variables. These individuals were randomized to compose the control group (CG) and the intervention group (GBS). The routine physical therapy was performed in both groups and in the GBS two daily sessions of up to 20 minutes of Breath Stacking technique were applied. To verify the effect of this intervention, before and after the protocol, patients underwent the following evaluations: algometry, cirtometry in the axillary line , umbilical line and the xiphoid process, ventilometry, spirometry and manovacuometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgical procedure that involves in an incision in the upper quadrants of the abdominal region.

Exclusion Criteria:

* Intolerance to the use of BS mask.
* Chronic obstructive pulmonary disease (COPD), Asthma, Chron's disease.
* Liver trauma severe with hemodynamic repercussions.
* Patients undergoing esophagectomy.
* Sepsis with complications postoperative hemodynamics.
* Need for surgical reintervention.
* Forwarded to Intensive Care Unit or need for mechanical ventilation after discharge from the anesthetic recovery.
* Cognitive dysfunction that makes it impossible to understand and execute evaluations and intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change from second postoperative day forced vital capacity (FVC) at 7th postoperative day or hospital discharge. | The change in FVC will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  The FVC will be evaluated as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
Change from second postoperative day tidal volume at 7th postoperative day or hospital discharge. | The change in tidal volume will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  Tidal volume will be obtained through the division of the minute volume by the respiratory rate.

SECONDARY OUTCOMES:
Heart rate | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day. This variable will also be measured before and after the first and last BS session.
  It will be evaluated with portable pulse oximeter.
Respiratory rate | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day. This variable will also be measured before and after the first and last BS session.
  The respiratory rate will be measured by the movements of the rib cage during respiratory cycles performed in one minute.
Blood pressure | These will be evaluated on the 2nd postoperative day and up to 7th postoperative day. These will also be measured before and after the first and last BS session.
  Systolic and diastolic blood pressure will be verified by a stethoscope and sphygmomanometer.
Peripheral oxygen saturation (SpO2) | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day. This variable will also be measured before and after the first and last BS session.
  It will be evaluated with portable pulse oximeter.
Painful perception in the surgical incision | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  The digital algometer will be used, which constitutes a dynamometer that exerts pressure with a rubber tip 1 cm in diameter on the skin, at a 90º angle, determining the pain threshold.
Thoracoabdominal mobility | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  The measuring tape will be positioned in three anatomical points: axillary fold, xiphoid appendix and umbilical line. The measurements will be performed at rest, after maximum inspiration and after maximum expiration.
Minute volume | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  To obtain the minute volume (MV), the patient will be instructed to inhale and exhale slowly using the Wright ® ventilometer (British Oxygen Company, London, England).
Forced expiratory volume in the first second (FEV1) | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  It will be evaluated as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
FEV1 / FVC ratio (FEV1 / FVC) | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  It will be evaluated as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
Peak expiratory flow (PEF) | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  It will be evaluated as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
Forced expiratory flow between 25 and 75% of the curve of FVC (FEF25-75) | It will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  It will be evaluated as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
Respiratory muscle strength | These will be evaluated on the 2nd postoperative day and up to 7th postoperative day.
  The maximal inspiratory and expiratory pressures will be evaluated with manovacuometer.
Degree of dyspnea | It will be evaluated before and after the application of the BS technique (therefore, only in GBS) on the 2nd postoperative day and up to 7th postoperative day.
  It will be evaluated using the modified Borg Scale, a vertical scale quantified from 0 to 10. Zero represents no symptoms and 10 represents the maximum of symptoms.
Rates of signs of respiratory discomfort (dizziness, tachypnea, sweating, use accessory musculature) | These will be evaluated before and after the application of the BS technique (therefore, only in GBS) on the 2nd postoperative day and up to 7th postoperative day.
  Evaluated through clinical inspection.
Rates of gastrointestinal symptoms (pain abdominal, nausea, vomiting) | These will be evaluated before and after the application of the BS technique (therefore, only in GBS) on the 2nd postoperative day and up to 7th postoperative day.
  Evaluated through clinical inspection.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Fernandes DDL, Righi NC, Rubin Neto LJ, Belle JM, Pippi CM, Ribas CZDM, Nichele LFI, Signori LU, Silva AMVD. Effects of the breath stacking technique after upper abdominal surgery: a randomized clinical trial. J Bras Pneumol. 2022 Mar 14;48(1):e20210280. doi: 10.36416/1806-3756/e20210280. eCollection 2022. PMID 35293484